CLINICAL TRIAL: NCT01254708
Title: A Pilot Study to Determine the Safety and Clinical Efficacy of Once-Weekly Inhaled AmBisome for the Prevention of Aspergillus Colonization in Lung Transplant Recipients
Brief Title: Safety and Efficacy Study of Inhaled AmBisome for Prevention of Aspergillus Colonization in Lung Transplant Recipients
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has been placed on hold due to unavailability of funding.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AGM201000428
Record Dates: First submitted 2010-11-22; First posted 2010-12-06 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Lung Transplant Recipient
MeSH Terms: interventions — liposomal amphotericin B

ARMS (2):
- Control (Active Comparator): Standard of care group. Medication as prescribed by the primary physician would be used by this group. Such medications might include azoles as voriconazole
  Interventions: Drug: Regular standard of care medication
- liposomal amphotericin B (AmBisome ®) (Experimental): Inhaled Liposomal preparation of Amphotericin B.
  Interventions: Drug: Ambisome ®

INTERVENTIONS:
Drug: Ambisome ® — liposomal amphotericin B
  Arms: liposomal amphotericin B (AmBisome ®)
Drug: Regular standard of care medication — Drug for this group is at the physician's discretion. Patients in this group receive the standard of care medication currently implemented at the Institution. Example would be voriconazole
  Arms: Control

SUMMARY:
Lung transplant recipients have the highest rate of Invasive Aspergillus (IA)infection among solid organ transplant recipients. The most important risk factor for the development of IA (which is associated with disease and death) is colonization of the organism in the respiratory tract.

Azoles are used to prevent the development of IA. Puffers containing antifungal medication can be used to treat the lungs without the need to worry about the medication interactions & side-effects in the blood. An example of this is the aerosolized amphotericin B. Its use is limited by the patients' tolerating this medication that may cause cough, nausea & contraction of the air pathways.

The lipid preparation is better tolerated and has longer dosing interval than inhaled amphotericin B. The investigators propose a pilot study to determine the long-term safety of inhaled AmBisome administration of drug and generate the preliminary data on the effectiveness of this drug to prevent aspergillus colonization.

DETAILED DESCRIPTION:
In this pilot study, our main aims are:

1. To determine the safety of once weekly Inhaled AmBisome prophylaxis in preventing the development of Aspergillus colonization in lung transplant recipients at one year of prophylaxis.
2. To generate the preliminary data on the efficacy of Inhaled AmBisome (Astellas) loading dose (1mg/kg/day for four days) initially followed by q weekly dosage to complete 1 year in lung transplant recipients as compared to no prophylaxis by assessing the rate of fungal colonization/infections between the groups.

ELIGIBILITY:
Inclusion Criteria:

1. Single or double lung transplant recipients who are at least one year out of transplantation.
2. Age >18yrs of age
3. Able to understand and complete informed consent.

Exclusion Criteria:

1. Pregnant woman or woman capable of bearing children, who will not perform urine pregnancy test.
2. Nursing mothers.
3. Subjects with hypersensitivity to Amphotericin deoxycholate or liposomal Amphotericin.
4. Subjects with a past history of bronchospasm associated with aerosol drug use.
5. Subjects with active bacterial or viral infection as defined by the current use of non-prophylactic antibiotic anti-viral medications.
6. Subjects treated with cytolytic medications (Campath /Thymoglobulin) within the last month.
7. Subjects with an FEV1< 30% Predicted or FVC% <30%.
8. Subjects requiring supplemental oxygen.
9. Receipt of Inhaled or IV Amphotericin B within last 30 days.
10. Subjects with known fungal infection as per MSG Criteria on therapy with antifungal drugs or diagnosed on the day of bronchoscopy.
11. Current use of azoles active against molds (Voriconazole, itraconazole, posaconazole) for the prophylaxis.
12. Serum creatinine > 150 mmol/L on the day of clinic visit.
13. Liver enzymes ALT/ AST/ Alkphos greater than two times upper limit of normal.
14. Concurrent intravenous aminoglycoside use.
15. Subjects with fever > 38.2°C.
16. Subjects on mechanical ventilation.
17. Expected survival less than 6 months.
18. Re-transplants and heart/lung transplant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function | Day 1 to 12 months
  Assess pulmonary function measurements i.e. changes in FEV1 (Forced Expiratory Volume 1), changes in FVC (Forced Vital Capacity) while receiving inhaled liposomal amphotericn B.
Symptoms | Day 1 to 12months
  Assess onset of symptoms including headache, dizziness and fatigue, fever, nausea, vomiting, wheezing, cough, shortness of breath, and taste preservation, while receiving inhaled liposomal amphotericin B
Renal or Hepatic dysfunction and Neutropenia | Day 1 to 12 months
  Assess the development of renal or hepatic dysfunction and neutropenia by measuring serum creatinine liver enzymes and white blood cells

SECONDARY OUTCOMES:
Presence of Invasive fungal infection | 1 year
  Measure the time in months from randomization of study participants to diagnosis of invasive fungal infection (proven or probable). Measure the time in months from randomization to death for study participants.
  Assessment of the quality of life at the baseline Month 0, 3, 6, 9 and 12 months based on responses to a questionnaire. These include responses to general questions to rate the level of emotions and the general well being of the study participants. These responses are rated as never, sometimes, often or always experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Husain, M.D M.Sc, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network/ Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Newman SP, Clarke SW. Therapeutic aerosols 1--physical and practical considerations. Thorax. 1983 Dec;38(12):881-6. doi: 10.1136/thx.38.12.881. No abstract available. PMID 6364439
- [Background] Barry PW, O'Callaghan C. Inhalational drug delivery from seven different spacer devices. Thorax. 1996 Aug;51(8):835-40. doi: 10.1136/thx.51.8.835. PMID 8795674
- [Background] Monforte V, Roman A, Gavalda J, Bravo C, Tenorio L, Ferrer A, Maestre J, Morell F. Nebulized amphotericin B prophylaxis for Aspergillus infection in lung transplantation: study of risk factors. J Heart Lung Transplant. 2001 Dec;20(12):1274-81. doi: 10.1016/s1053-2498(01)00364-3. PMID 11744410
- [Background] Calvo V, Borro JM, Morales P, Morcillo A, Vicente R, Tarrazona V, Paris F. Antifungal prophylaxis during the early postoperative period of lung transplantation. Valencia Lung Transplant Group. Chest. 1999 May;115(5):1301-4. doi: 10.1378/chest.115.5.1301. PMID 10334143
- [Background] Cicogna CE, White MH, Bernard EM, Ishimura T, Sun M, Tong WP, Armstrong D. Efficacy of prophylactic aerosol amphotericin B lipid complex in a rat model of pulmonary aspergillosis. Antimicrob Agents Chemother. 1997 Feb;41(2):259-61. doi: 10.1128/AAC.41.2.259. PMID 9021176
- [Background] Drew RH, Dodds Ashley E, Benjamin DK Jr, Duane Davis R, Palmer SM, Perfect JR. Comparative safety of amphotericin B lipid complex and amphotericin B deoxycholate as aerosolized antifungal prophylaxis in lung-transplant recipients. Transplantation. 2004 Jan 27;77(2):232-7. doi: 10.1097/01.TP.0000101516.08327.A9. PMID 14742987
- [Background] Palmer SM, Drew RH, Whitehouse JD, Tapson VF, Davis RD, McConnell RR, Kanj SS, Perfect JR. Safety of aerosolized amphotericin B lipid complex in lung transplant recipients. Transplantation. 2001 Aug 15;72(3):545-8. doi: 10.1097/00007890-200108150-00036. PMID 11502995
- [Background] Schwartz S, Behre G, Heinemann V, Wandt H, Schilling E, Arning M, Trittin A, Kern WV, Boenisch O, Bosse D, Lenz K, Ludwig WD, Hiddemann W, Siegert W, Beyer J. Aerosolized amphotericin B inhalations as prophylaxis of invasive aspergillus infections during prolonged neutropenia: results of a prospective randomized multicenter trial. Blood. 1999 Jun 1;93(11):3654-61. PMID 10339471
- [Background] Corcoran TE, Venkataramanan R, Mihelc KM, Marcinkowski AL, Ou J, McCook BM, Weber L, Carey ME, Paterson DL, Pilewski JM, McCurry KR, Husain S. Aerosol deposition of lipid complex amphotericin-B (Abelcet) in lung transplant recipients. Am J Transplant. 2006 Nov;6(11):2765-73. doi: 10.1111/j.1600-6143.2006.01529.x. PMID 17049064
- [Background] Monforte V, Roman A, Gavalda J, Lopez R, Pou L, Simo M, Aguade S, Soriano B, Bravo C, Morell F. Nebulized amphotericin B concentration and distribution in the respiratory tract of lung-transplanted patients. Transplantation. 2003 May 15;75(9):1571-4. doi: 10.1097/01.TP.0000054233.60100.7A. PMID 12792517